CLINICAL TRIAL: NCT06468501
Title: Socioeconomic Position and the Effectiveness of Price Changes Based on Healthier and Less Healthy Food on Food Selection in a Simulated Out of Home Food Delivery App: a Randomised Controlled Trial
Brief Title: SEP and the Impact of Price on Food Selection in a Simulated Food Delivery App
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Principal Investigator, Eric Robinson, Professor, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Food Delivery Study
Record Dates: First submitted 2024-06-11; First posted 2024-06-21 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-06

CONDITIONS: Food Selection; Healthy Eating; Eating Behavior
MeSH Terms: conditions — Food Preferences; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: The design is a randomised controlled trial, with 4 (interventions) x 2 (high vs low SEP) between-subject conditions.
Who Masked: Participant, Investigator
Masking Description: This study will be double-blinded, which means that both the participants and the researchers are not aware in which treatment group participants are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Price reduction on healthier foods (Experimental): * Price reduction of 10% for healthier dishes (based on a score of less than 4 on the UK Nutrient Profile Model (NPM))
  * Existing price structure for less healthy dishes (based on a score of 4 or higher on the UK NPM)
  Interventions: Behavioral: Price reduction on healthier foods
- Price increase to less healthy foods (Experimental): * Price increase of 10% for less healthy dishes (based on a score of less than 4 on the UK NPM)
  * Existing price structure for healthier dishes (based on a score of 4 or higher on the UK NPM)
  Interventions: Behavioral: Price increase to less healthy foods
- Combination of price reduction to healthier foods and price increase to less healthy foods (Experimental): * Price reduction of 10% for healthier dishes (based on a score of less than 4 on the UK NPM)
  * Price increase of 10% for less healthy dishes (based on a score of 4 or higher on the UK NPM)
  Interventions: Behavioral: Combination of price reduction on healthier foods and price increase on less healthy foods
- Existing price structure (control) (Placebo Comparator): - No changes in prices
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Price reduction on healthier foods — Price reduction (10%) on healthier foods based on the UK NPM
  Arms: Price reduction on healthier foods
Behavioral: Price increase to less healthy foods — Price increase (10%) on less healthy foods based on the UK NPM
  Arms: Price increase to less healthy foods
Behavioral: Combination of price reduction on healthier foods and price increase on less healthy foods — Combination of price reduction (10%) on healthier foods based on the UK NPM and price increase (10%) on less healthy foods based on the UK NPM
  Arms: Combination of price reduction to healthier foods and price increase to less healthy foods
Behavioral: Control — Existing price structure
  Arms: Existing price structure (control)

SUMMARY:
The goal of this randomised controlled trial is to compare taxation with subsidies to encourage healthier food choices in the out-of-home food sector. Participants will be asked to make hypothetical food choices in an online simulation study of a delivery app. Participants will be randomised into four different intervention groups:

1. Price reduction (10%) on healthier foods
2. Price increase (10%) to less healthy foods
3. A combination of price reduction to healthier foods and price increase to less healthy foods
4. Existing price structure (i.e. control group)

The investigators will further examine effectiveness of these fiscal policies on healthy eating by socioeconomic position to understand whether these policies are equitable.

ELIGIBILITY:
Inclusion Criteria:

* Currently reside in the United Kingdom
* Over the age of 18 years
* Order take-away food for delivery at least once a month
* Can complete the study on a laptop or desktop

Exclusion Criteria:

* Any major dietary restrictions (vegan, dairy/lactose-free, gluten-free) or allergies (dairy, eggs, nuts, soy, wheat) that would limit the number of dishes they could choose in the meal selection task

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3464 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Healthier vs less healthy main meals ordered based on the Nutrient Profiling Model and total energy (kcal) | immediately after food choice
  Healthier vs less healthy main meals ordered
Total energy (kcal) ordered | immediately after food choice
  The total energy content of the total hypothetical food order

SECONDARY OUTCOMES:
Proportion of selecting healthier vs less healthy meal items of the total food order based on the Nutrient Profiling Model and total energy (kcal) | immediately after food choice
  Proportion of selecting healthier vs less healthy meal items of the total hypothetical food order
Total fat, saturated fat, salt and sugar ordered | immediately after food choice
  Total fat, saturated fat, salt and sugar of total hypothetical food order

CONTACTS AND LOCATIONS:
Overall Officials: Eric Robinson, PhD, Principal Investigator — University of Liverpool
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Study data (anonymised) will be shared on the Open Science Framework (OSF)
Supporting Information: Study Protocol, SAP
Time Frame: On publication, indefinitely
Access Criteria: Open website